CLINICAL TRIAL: NCT00409799
Title: A Phase 2 Randomized, Controlled, Open-label (Dose-blinded), Multi-center, Dose-finding Study of the Safety and Efficacy of I-0401 in the Treatment of Patients With Fractures of the Tibial Plateau Requiring Grafting.
Brief Title: Safety and Efficacy of I 0401 in the Treatment of Tibial Plateau Fractures Requiring Grafting
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kuros Biosurgery AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CS I-040101/02
Record Dates: First submitted 2006-12-08; First posted 2006-12-11 (Estimated); Last update posted 2012-03-16 (Estimated); Status verified 2012-03

CONDITIONS: Tibia Plateau Fractures
Keywords: Bone graft substitute; Promotion of bone healing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Experimental - high dose
  Interventions: Drug: I-0401 (a new bone graft substitute)
- 2 (Experimental): Experimental - low dose
  Interventions: Drug: I-0401 (a new bone graft substitute)
- 3 (Active Comparator): Autograft
  Interventions: Drug: I-0401 (a new bone graft substitute)

INTERVENTIONS:
Drug: I-0401 (a new bone graft substitute) — 1 time application

SUMMARY:
For certain tibial plateau fractures the bone is compressed due to the force acting on the tibia during the accident. The void provoked by the compression of the bone is filled with an appropriate filling material and the fracture is fixated. I 0401 is a new bone graft substitute that has shown capacities to promote bone-healing. This study will test the safety and efficacy of I 0401 in the treatment of patients with tibial plateau fractures requiring grafting.

ELIGIBILITY:
Inclusion Criteria:

* Radiological evidence of a tibial plateau fracture requiring grafting
* Females of child-bearing potential must be willing to undergo a pregnancy test (urine) prior to treatment start (at screening).

Exclusion Criteria:

* Concomitant ipsilateral fractures of the limb other than the fracture of the tibial plateau.
* Active or past history of malignant tumor.
* Evidence of systemic or localized infection at time of surgery.
* Pregnant or lactating females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2006-11; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Radiographic Images | All Follow-Up Visits

SECONDARY OUTCOMES:
Clinical assessments of the fracture site | All Follow-Up Visits
Blood parameters | All Follow-Up Visits
Vital signs | At several Follow-Up visits
Questionnaires of Life | All Follow-Up Visits
Pharmacoeconomic evaluation | All Follow-Up Visits

CONTACTS AND LOCATIONS:
Overall Officials: Peter Messmer, MD, Principal Investigator — Zurich University Hospital, Zurich, Switzerland
Locations (45):
- Australia (3):
  - Gold Coast Hospital (49), Gold Coast, Queensland
  - Princess Alexandra Hospital (45), Woollongabba, Queensland
  - Royal Adelaide Hospital (48), Adelaide, South Australia
- France (4):
  - Hopital La Cavale Blanche (19), Brest
  - Hôpital de Dunkerque (30), Dunkirk
  - Hôpital Central de Nancy (05), Nancy
  - Hôpital Charles Nicolle (15), Rouen
- Germany (8):
  - Charite, Campus Virchow Klinikum (03), Berlin
  - Berufsgenossenschaftliche Unfallklinik Bochum/Duisburg (11), Duisburg
  - Uniklinik Göttingen (22), Göttingen
  - Med. Hochschule Hannover (06), Hanover
  - Universitätsklinikum Schleswig-Holstein (40), Kiel
  - St.-Josef-Krankenhaus (12), Linnich
  - Chirurgische Klinik der LMU (50), München
  - Universitätsklinikum Münster (39), Münster
- Hungary (5):
  - Fövarosi Önkormanyzat Karolyi Sandor Korhaz es Rendelointezet (21), Budapest
  - Fövarosi Önkormanyzat Peterfy Sandor utcai Korhaz-Rendelöinezet es Baleseti Központ (20), Budapest
  - Fovárosi Önkormányzat Szent János Kórháza és Észak (54), Budapest
  - Petz Alandar County Teaching Hospital (55), Győr
  - Szegedi Egyetem AOK Kari Gyogyszertar (27), Szeged
- Italy (5):
  - Istituti Ortopedici Rizzoli (13), Bologna
  - Fondazione Istituto San Raffaele G. Giglio di Cefalù (16), Cefalù
  - A.O. Universitaria San Martino (33), Genova
  - Università degli Studi di Roma "Tor Vergata" (10), Roma
  - A.O. San Giovanni Oddolorata (14), Roma
- Poland (6):
  - Klinika i Oddzial Kliniczny - Ortopedii i Traumatologii (36), Krakow
  - Oddzial Chirurgii Ortopedyczno-Urazowej - Wojewodzki Szpital Specjalistyczny (58), Lodz
  - SPZOZ Wojewodzki - Specjalistyczny Szpital Chirurgii Urazowej (35), Piekary Śląskie
  - Katedra i Klinika Ortopedii - Traumatologii PAM (34), Szczecin
  - Wojskowy Instytut Medyczny - Centralny Szpital Kliniczny MON (60), Warsaw
  - Katedra I Klinika Ortopedii AM (29), Warsaw
- Spain (5):
  - Hospital Universitario de la Princesa (18), Madrid
  - Hospital FREMAP Majadahonda (17), Madrid
  - Hospital Universitario Virgen de la Victoria (51), Málaga
  - Hospital FREMAP Sevilla (32), Seville
  - Hospital Universitario La Fe (07), Valencia
- Switzerland (5):
  - Zurich University Hospital (01), Zurich, Canton Zurich
  - Universitätsspital Basel (24), Basel
  - Kantonsspital Bruderholz (25), Bruderholz
  - CHUV Lausanne (02), Lausanne
  - Kantonsspital Luzern (26), Lucerne
- United Kingdom (4):
  - Leeds General Infirmary (04), Leeds, West Yorkshire
  - N. Bristol NHS Trust + Univ. of Bristol (52), Bristol
  - University Hospital of Wales (31), Cardiff
  - Norfolk and Norwich University Hospital (44), Norwich

REFERENCES:
- [Derived] Smith TO, Casey L, McNamara IR, Hing CB. Surgical fixation methods for tibial plateau fractures. Cochrane Database Syst Rev. 2024 Aug 22;8(8):CD009679. doi: 10.1002/14651858.CD009679.pub3. PMID 39171616